CLINICAL TRIAL: NCT05993923
Title: Impact of a Multidisciplinary Approach in the Perioperative Geriatrics Unit on Functional Status of Patients Aged 70 and Over Operated on for Colorectal Cancer. Randomized Open-label Controlled Study
Brief Title: Impact of a Multidisciplinary Approach in the Perioperative Geriatrics Unit on Functional Status of Patients Aged 70 and Over Operated on for Colorectal Cancer
Acronym: DIGER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NIMAO/2022-2/CL-01
Record Dates: First submitted 2023-06-13; First posted 2023-08-15 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2024-12

CONDITIONS: Colorectal Cancer; Surgery
Keywords: Elderly; Geriatric Unit; Postoperative
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Classical management in the digestive surgery department
- GPOU group (Experimental): Treatment is carried out in Peri-Operative Geriatrics Unit to optimize specific geriatric care
  Interventions: Other: GPOU

INTERVENTIONS:
Other: GPOU — Intervention upstream of the perioperative management according to the nutritional grade. Grade 4 Nutrition patients will be hospitalized earlier, i.e. 10 to 15 days before surgery for the start of artificial nutrition. A temporary return home can be organized with the supervision of a service provider until a second admission for surgical management. Grade 2 Nutrition patients will be called 24 to 48 hours before the surgical procedure.
  Anticipation of discharge at admittance Early mobilization Comorbidity management Prevention of iatrogenia Management of geriatric frailties Daily medical and paramedical assessment Detailed discharge report
  Arms: GPOU group

SUMMARY:
Health establishments encourage the development of specific care pathways for the elderly by supporting Geriatric Peri-Operative Units (GPOU). Indeed, this shared care model has shown a clear reduction in mortality and the number of re-hospitalizations in patients 6 months after their care. The multidisciplinary approach of global management of the patient in the perioperative period aims to reduce surgical stress as well as the rapid restoration of previous physical and psychic abilities. Colorectal surgery, the main treatment for stage I to III colon cancer, is a morbid surgery. Despite numerous efficacy data on improved rehabilitation after colorectal surgery, care programs are not specific to the geriatric population and geriatric assessment criteria to describe the functional status of patients are not commonly used. The study investigators wish to evaluate the impact of GPOU treatment following colorectal surgery, on the evolution of several clinical parameters such as: functional status, morbidity mortality, quality of life, and lifestyle. The study investigators hypothesize that management in the GPOU for colorectal cancer surgery in patients aged 70 and over will improve functional status at 3 months, in comparison with traditional management. The proposed intervention should also lead to an improvement in patient satisfaction with care, complications and re-hospitalizations, nutritional status, lifestyle and patient survival.

ELIGIBILITY:
Inclusion Criteria:

* The patient or their representative must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* Diagnosis of proven colorectal cancer.
* Patient to benefit from scheduled colorectal surgery at the University Hospital of Nîmes validated in digestive surgery SPC after oncogeriatric evaluation.
* Surgical act: resection with anastomosis in one step.

Exclusion Criteria:

* Interventional RIPH patient defined as category 1 if there is interference with the primary endpoint
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-09-26 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Change in functional status after colorectal cancer surgery between groups | Baseline and Month 3
  Instrumental Activities of Daily Living (IADL) score (score 0-8)

SECONDARY OUTCOMES:
Change in functional status between groups | Baseline and Month 6
  Instrumental Activities of Daily Living (IADL) score (score 0-8)
Change in basic functional status between groups | Baseline, hospital discharge (an average of 10 days), Month 3, and Month 6
  Katz index of independence in Activities of Daily Living scale (ADL) (score 0-6)
Change in patient motor ability between groups | Baseline, Month 3
  Time Up and Go test (Score 0-3 for each item, time in seconds)
Patient satisfaction with care between groups | Hospital discharge (an average of 10 days)
  EORTC SATisfaction with IN-PATient cancer care (IN-PATSAT) 32 questionnaire (Score 32-160)
Length of hospital stay between groups | Hospital discharge (an average of 10 days)
  Days
The number of medical complications during hospitalization between groups | Hospital discharge (an average of 10 days)
  Number of following events: diabetes decompensation, cardiorespiratory decompensation, pulmonary and urinary infections, acute renal failure, anemia. Aggravation of: confusion, pelvic exoneration disorders, fall, bedsores.
The distribution of surgical complications between groups | Hospital discharge (an average of 10 days)
  Gravity of surgical complications according to the Clavien Dindo classification
The distribution of surgical complications between groups | Month 1
  Gravity of surgical complications according to the Clavien Dindo classification
Destination of patients on discharge from hospital between groups | Hospital discharge (an average of 10 days)
  Classified as: home / nursing home or institutionalization / transfer to Aftercare and Rehabilitation / transfer to another service / none (death during hospitalization).
The change in the patient's weight between groups | Baseline and Month 3
  Percent change in Kg
Patient quality of life between groups | Month 3
  EORTC-QLQ-C30 questionnaire score (Score 0-100)
Patient quality of life between groups | Month 6
  EORTC-QLQ-C30 questionnaire score (Score 0-100)
Change in the patient's place of abode between groups | Month 1, Month 3 and Month 6
  Rate (%) of patients living at home/in nursing home/residential home
Overall survival between groups. | Month 1
  Percentage of immediate mortality (during the hospital stay)
Overall survival between groups. | Month 3
  Percentage of immediate mortality (during the hospital stay)
Overall survival between groups. | Month 6
  Percentage of immediate mortality (during the hospital stay)
The rate of early unscheduled re-hospitalizations or admissions to the emergency department between groups | Month 1
  Re-hospitalization in the month following discharge from hospital: yes/no.

CONTACTS AND LOCATIONS:
Overall Officials: Coralie Labarias, Principal Investigator — CHU de Nimes
Locations (2):
- France (2):
  - Coralie LABARIAS, Nîmes, France
  - CHU de Nîmes, Nîmes